CLINICAL TRIAL: NCT00050557
Title: Family Psychoeducation: Efficacy in Child Mood Disorders
Brief Title: Family Psychoeducation for Children With Mood Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mary Fristad (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Mary Fristad, Professor, Psychiatry, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH061512 (NIH); R01MH061512 (NIH); DSIR CT-S
Record Dates: First submitted 2002-12-13; First posted 2002-12-16 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Mood Disorders
MeSH Terms: conditions — Mood Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive immediate Multi-Family Psychoeducation Group treatment and ongoing treatment as usual
  Interventions: Behavioral: Multifamily Psychoeducation Group (MFPG); Behavioral: Treatment as usual (TAU)
- 2 (Active Comparator): Participants will receive treatment as usual and waitlist Multi-Family Psychoeducation Group treatment
  Interventions: Behavioral: Multifamily Psychoeducation Group (MFPG); Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Multifamily Psychoeducation Group (MFPG) — MFPG will include 8 weekly 90-minute group therapy sessions.
Behavioral: Treatment as usual (TAU) — Participants will receive standard care for mood disorders.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a Multifamily Psychoeducation Group for the families of children with mood disorders.

DETAILED DESCRIPTION:
Mood disorders among youth are a major health concern. Existing mood disorder studies focus on adults, and studies that focus on effective intervention strategies for youth with mood disorders are needed. This 8-session study is an adjunct to ongoing medication management and individual and family psychotherapy for children with mood disorders.

In this study, parents learn about mood disorders, their treatments, and how to work effectively with mental health and school systems. Parents also practice problem-solving and communication skills for symptom management. Children learn about mood disorders and their treatments, including basic cognitive-behavioral principles. Children also learn and practice anger management, problem-solving, and communication skills.

Patients and their families are randomly assigned to 1 of 2 groups. The first group receives 8 sessions of psychoeducation plus treatment as usual (TAU). The second group is a wait-list control in which participants receive only TAU. Patients and caregivers undergo a variety of interviews, tests, and behavioral observations throughout the study. Anxiety, depression, psychosocial stressors, manic symptoms, and children's experiences with psychotropic medications and with treatment or service providers are assessed. Caregivers, teachers, and family friends undergo interviews and make observations of the patient's level of support, general appearance and behavior, and overall functional capacity. The extent to which caregivers agree on the need for treatment and the extent of caregivers' knowledge of mood disorders is also assessed. Assessments occur at 3, 6, 12, 15, and 18 months after study enrollment. A comprehensive assessment is conducted at study entry and 1 year later.

ELIGIBILITY:
Inclusion criteria:

* Major depressive disorder, dysthymic disorder, or bipolar disorder (Type I or II)
* IQ greater than 70
* At least one parent/caregiver willing to participate in the study
* Able to attend six or more of the eight treatment sessions with at least 1 parent

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2001-07; Primary Completion 2006-09 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Mood Severity Index | Measured at Months 6 and 12

SECONDARY OUTCOMES:
Rage Index (MRS irritability + disruptive-aggressive items) | Measured at Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Mary A. Fristad, PhD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Derived] Boylan K, Macpherson HA, Fristad MA. Examination of disruptive behavior outcomes and moderation in a randomized psychotherapy trial for mood disorders. J Am Acad Child Adolesc Psychiatry. 2013 Jul;52(7):699-708. doi: 10.1016/j.jaac.2013.04.014. PMID 23800483
- [Derived] Fristad MA, Verducci JS, Walters K, Young ME. Impact of multifamily psychoeducational psychotherapy in treating children aged 8 to 12 years with mood disorders. Arch Gen Psychiatry. 2009 Sep;66(9):1013-21. doi: 10.1001/archgenpsychiatry.2009.112. PMID 19736358